CLINICAL TRIAL: NCT00710606
Title: Comparison of Serum Contraceptive Hormone Levels Between Normal Weight and Obese Users of the NuvaRing®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Organon (Industry)
Responsible Party: Principal Investigator, Carolyn L. Westhoff, Director of Family Planning and Preventive Services Division, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: AAAC8127
Record Dates: First submitted 2008-07-01; First posted 2008-07-04 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Pharmacokinetics
Keywords: contraceptive ring; obesity; pharmacokinetics; pharmacodynamics; Pharmacokinetics of the contraceptive ring in obese women.
MeSH Terms: conditions — Obesity | interventions — NuvaRing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1- Obese Women /Nuvaring (Experimental): Obese subjects (BMI 30-39.9)received two contraceptive hormonal rings. During the second cycle of ring use, subjects returned to the study site for serial serum hormone measurements and transvaginal ultrasound twice weekly during four weeks of continuous use.
  Interventions: Drug: NuvaRing
- 2- Normal Weight / Nuvaring (Active Comparator): Normal weight subjects (BMI 19-24.9) received two contraceptive hormonal rings. During the second cycle of ring use, subjects returned to the study site for serial serum hormone measurements and transvaginal ultrasound twice weekly during four weeks of continuous use.
  Interventions: Drug: NuvaRing

INTERVENTIONS:
Drug: NuvaRing — Obese subjects (BMI 30-39.9) will receive two contraceptive hormonal rings. During the second cycle of ring use, subjects will return to the study site for serial serum hormone measurements and transvaginal ultrasound twice weekly during four weeks of continuous use.
  Arms: 1- Obese Women /Nuvaring
Drug: NuvaRing — Normal weight subjects will also receive two contraceptive hormonal rings. During the second cycle of ring use, subjects will return to the study site for serial serum hormone measurements and transvaginal ultrasound twice weekly during four weeks of continuous use.
  Arms: 2- Normal Weight / Nuvaring

SUMMARY:
There are over 60 million women of reproductive age in the U.S. and a majority of these women qualify as overweight or obese. Evidence suggests that there is an association between increased body weight and decreased contraceptive efficacy. Studies with the combined hormonal contraceptive patch (Evra®) and the subdermal contraceptive implant (Norplant®) demonstrate higher failure rates in heavier versus lighter women.

Weight related differences in the effectiveness of NuvaRing® need further study. A single secondary analysis of pooled data from Phase III clinical trials of NuvaRing® noted no difference in pregnancy rates among women in the highest weight decile (>166#) versus the rest of the study population using the ring. (Westhoff, 2005) The finding of no difference, however, was influenced by too few obese subjects in the analysis which contributed to wide confidence limits. Additional studies are needed to explore how well the contraceptive ring functions to maintain effective serum steroid concentrations to suppress ovarian activity in obese women.

This investigation focused on evaluating mean serum concentrations of hormones released in obese and normal weight women using the NuvaRing® . This study was a prospective clinical trial. Normal weight women are defined as women with a BMI 19-24.9 and obese women are those with a BMI 30-39.9. We recruited forty adult women interested in initiating the combined hormonal contraceptive ring to two months of use to complete analysis of at least 34 subjects (17 normal weight, 17 obese). We compared mean serum concentrations of ethinyl estradiol (E2) and etonogestrel (ENG) along with additional markers for ovarian suppression. These markers included sonographic evidence of follicular development and ovulation as well as circulating E2 levels which strongly correlate with follicular development and endometrial proliferation during the second month of NuvaRing® use. Assessment of these parameters will translated to understanding contraceptive-mediated suppression of ovarian function in these two groups. Subjects also logged patterns of ring use and bleeding patterns during the study period.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 yo
* Meet BMI requirements
* Weight stable
* English speaking
* Desire contraception
* History of regular menses with normal uterus and ovaries
* Medically eligible for combined hormonal contraception
* Tolerates phlebotomy/TVS

Exclusion Criteria:

* Exclusion:
* Heavy smokers
* Users of medications that alter hormone levels

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Westhoff, MD, MSc, Principal Investigator — Columbia University
Locations (1):
- Division of Family Planning and Preventive Services, New York, New York, United States

REFERENCES:
- [Background] Gu S, Sivin I, Du M, Zhang L, Ying L, Meng F, Wu S, Wang P, Gao Y, He X, et al. Effectiveness of Norplant implants through seven years: a large-scale study in China. Contraception. 1995 Aug;52(2):99-103. doi: 10.1016/s0010-7824(95)00141-7. PMID 8536454
- [Background] Sivin I, Lahteenmaki P, Mishell DR Jr, Alvarez F, Diaz S, Ranta S, Grozinger C, Lacarra M, Brache V, Pavez M, Nash H, Stern J. First week drug concentrations in women with levonorgestrel rod or Norplant capsule implants. Contraception. 1997 Nov;56(5):317-21. doi: 10.1016/s0010-7824(97)00153-4. PMID 9437561
- [Background] Sivin I, Wan L, Ranta S, Alvarez F, Brache V, Mishell DR Jr, Darney P, Biswas A, Diaz S, Kiriwat O, Anant MP, Klaisle C, Pavez M, Schechter J. Levonorgestrel concentrations during 7 years of continuous use of Jadelle contraceptive implants. Contraception. 2001 Jul;64(1):43-9. doi: 10.1016/s0010-7824(01)00226-8. PMID 11535213
- [Background] Smallwood GH, Meador ML, Lenihan JP, Shangold GA, Fisher AC, Creasy GW; ORTHO EVRA/EVRA 002 Study Group. Efficacy and safety of a transdermal contraceptive system. Obstet Gynecol. 2001 Nov;98(5 Pt 1):799-805. doi: 10.1016/s0029-7844(01)01534-4. PMID 11704172
- [Background] Westhoff, C. Higher body weight does not affect NuvaRing's efficacy. Obstet Gynecol 2005; 104: 56S.
- [Background] Zieman M, Guillebaud J, Weisberg E, Shangold GA, Fisher AC, Creasy GW. Contraceptive efficacy and cycle control with the Ortho Evra/Evra transdermal system: the analysis of pooled data. Fertil Steril. 2002 Feb;77(2 Suppl 2):S13-8. doi: 10.1016/s0015-0282(01)03275-7. PMID 11849631

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled during the months of June-September 2008.
Groups:
- Obese Subjects: Obese subjects (BMI 30-39.9) received two contraceptive hormonal rings. During the second cycle of ring use, subjects returned to the study site for serial serum hormone measurements and transvaginal ultrasound twice weekly during four weeks of continuous use.
- Normal Weight Subjects: Normal weight subjects (BMI 19-24.9) received two contraceptive hormonal rings. During the second cycle of ring use, subjects returned to the study site for serial serum hormone measurements and transvaginal ultrasound twice weekly during four weeks of continuous use.
Period: Overall Study
Arm/Group | Obese Subjects | Normal Weight Subjects
Started | 20 | 20
Completed | 20 | 18
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Obese Subjects: Obese subjects (BMI 30-39.9)
- Normal Weight Subjects: Normal weight subjects (BMI 19-24.9)
- Total: Total of all reporting groups
Arm/Group | Obese Subjects | Normal Weight Subjects | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.5 (3.2) | 26.0 (3.6) | 25.8 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Mean Serum Concentrations of Etonogestrel and Ethinyl Estradiol
Description: Serum concentrations were obtained from thirty-seven women completed follow-up.
Time Frame: Measurements at Week 3 and Week 6 continuous ring use
Population: 17 participants in each group was planned a priori to have 80% power to identify a one standard deviation difference in the mean serum levels of the contraceptive hormones. We enrolled 40 women, 2 withdrew prior to the study cycle. We excluded one woman due to removal of the CVR during the study cycle leaving 18 normal weight and 19 obese women.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/L
Groups:
- Normal Weight; Obese: Women of normal weight and obese received two contraceptive rings. During the second cycle of ring use, subject returned to the study site for serial serum hormone measurements and transvaginal ultrasound twice weekly during four weeks of continuous use.
Arm/Group | Normal Weight | Obese
Number analyzed (Participants) | 18 | 19
ng/L
  Etonogesterel (ENG) Week 3 | 1275 [1116 to 1457] | 1240 [1041 to 1477]
  Ethinyl Estradiol (EE) Week 3 | 21.9 [17.9 to 26.6] | 14.8 [12.7 to 17.3]
  Etonogesterel (ENG) Week 6 | 1063 [730 to 1548] | 1096 [730 to 1646]
  Ethinyl Estradiol (EE) Week 6 | 16.2 [10.1 to 25.8] | 12.5 [8.1 to 19.5]

2. Secondary Outcome: Number of Participants Achieving a Maximum Follicle Diameter > 13mm During the 3 Weeks of Follow-up
Description: Follicular development was minimal in both groups, with only five women achieving a maximum follicle diameter > 13mm at any time during the 3 weeks of follow-up (3 normal weight and 2 obese women).
Time Frame: continuous ring use, an average of 3 weeks
Population: as for outcome 1
Measure: Number; unit: Participant w/follicular diameter >=13mm
Arm/Group | Obese Subjects | Normal Weight Subjects
Number analyzed (Participants) | 19 | 18
Participant w/follicular diameter >=13mm | 2 | 3

3. Secondary Outcome: Mean Endometrial Proliferation
Description: The mean endometrial proliferation from week 1, week 2 and week3
Time Frame: Transvaginal ultrasound measurements of endometrial proliferation will be completed over continuous ring use, an average of 3 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Obese Subjects | Normal Weight Subjects
Number analyzed (Participants) | 19 | 18
millimeters | 4.7 (1.8) | 3.9 (1.6)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Obese Subjects | Normal Weight Subjects
Serious Adverse Events (participants affected / at risk) | 0/20 | 2/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obese Subjects (N=20) | Normal Weight Subjects (N=20)
fractured pelvis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) — deep vein thrombosis of lower extremity during treatment. additional risk fact was long haul air travel

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No